CLINICAL TRIAL: NCT01688765
Title: Longitudinal Multimodal Neuroimaging Studies in Patients With First Episode Psychosis
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Dost Ongur, M.D, PhD, Clinical Director, Mclean Hospital
Other Study IDs: 2012P001796
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Psychotic Disorders
Keywords: Schizophrenia; Schizoaffective disorder; Bipolar disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Episode Psychosis Patients: Individuals experiencing a first episode of psychosis
  Interventions: Other: Observational
- Healthy Controls: Psychiatrically healthy individuals
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
The purpose of this study is to investigate the structural, functional and chemical brain abnormalities in patients with first episode psychosis and assess the evolution of these abnormalities during the course of the disease.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the structural, functional and chemical brain abnormalities in patients with first episode psychosis and assess the evolution of these abnormalities during the course of the disease.

The study design is case-control, there are no interventions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of first episode of a psychotic disorder
* Healthy controls with no psychiatric disorder history

Exclusion Criteria:

* Significant neurological or medical illness history
* Ages <18 or >45

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: First episode psychosis patients Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States